CLINICAL TRIAL: NCT03739008
Title: Reversible Cerebral Vasoconstriction Syndrome With Concomitant Transient Global Amnesia : a Serie of 3 Cases Report
Brief Title: Reversible Cerebral Vasoconstriction Syndrome With Concomitant Transient Global Amnesia
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0423
Record Dates: First submitted 2018-11-09; First posted 2018-11-13 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2018-11

CONDITIONS: Transient Global Amnesia; Reversible Vasoconstriction Syndrome
Keywords: Thunderclap headache
MeSH Terms: conditions — Amnesia, Transient Global; Headache Disorders, Primary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Reversible cerebral vasoconstriction syndrome (RCVS) is characterized by severe, unusual headaches associated with multifocal segmental vasoconstriction of the intracerebral arteries. In addition to headache, focal neurological deficit and/or seizures are quite frequently described, but anterograde amnesia seems to but extremely rare. Indeed, to date, only one case of RCVS associated with transient global amnesia (TGA) has been published. In case of an atypical presentation of TG, associated with brutal headaches, it is important not to ignore an assocation with RCVS because management, treatment, evolution and prognosis are different. Indeed, TGA is a monophasic phenomenon of less than 24 hours duration, without associated complications, which does not require any particular treatment. On the other hand, RCVS, although most often of excellent prognosis, can have severe complications such as intracerebral hemorrhage, subarachnoid hemorrhage, posterior reversible encephalopathy syndrome and cerebral infarction. In order to limit headaches and potential complications, RCVS require special management, including symptomatic treatments for headaches, complete rest, removal of precipitin factors and introduction of calcium channel blockers for a few weeks.

This study aim to described three cases of patient who presented with concomitant TGA and RCVS, and to discuss pathogenic mechanism which may be similar in both these pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a proven or probable RCVS concomitant with certain transient global amnesia

Exclusion Criteria:

* Not proven transient global amnesia, not proven or possible RCVS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a proven or probable RCVS concomittant with certain transient global amnesia in the Neurology department of Gui de Chauliac and Lariboisière hospitals
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2018-11-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of concomitant TGA and proven RCVS | 1 day
  Occurrence of concomitant transient global amnesia (TGA) and proven Reversible cerebral vasoconstriction syndrome (RCVS)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Gaillard, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC